# ClinicalTrials.gov Data Entry Cover Sheet

**Protocol ID:** 21985IRB **Clinical Trials.gov ID:** NCT05521906

**Project Title**: Evaluation of PRYSHM for LGBTQIA2S+ Youth

Principal Investigator: Katie M. Edwards, PhD, University of Nebraska-Lincoln

Document Date: 3/20/2020

# Section 4 - Protocol Synopsis (Study 1)

#### 4.1. Brief Summary

Alcohol use (AU) and dating violence (DV) are serious public health problems in the U.S. that disproportionately impact LGBTQ+ youth. To date there is no comprehensive prevention program that concurrently addresses AU and DV among LGBTQ+ youth, which is sorely needed given the preliminary data suggest that traditional prevention programs do not work as well for this population. The purpose of the proposed study is to develop and evaluate an innovative, online-delivered program for LGBTQ+ youth that seeks to prevent AU and DV.

#### 4.2. Study Design

#### 4.2.a. Narrative Study Description

Following the initial creation of the online prevention program, we will conduct an online pilot trial to determine acceptability and feasibility to inform further refinement. Next, we will conduct a pilot RCT in which LGBTQ+ youth are recruited and randomly assigned to the intervention group (N=100) or to the wait list control group (N=100). Pre-, immediate, and three-month follow-up surveys will be used to assess the initial efficacy of the intervention in reducing AU and DV along with a number of other intermediary and secondary outcomes. Program observations as well as exit interviews will be used to further refine the intervention.

## 4.2.b. Primary Purpose

Prevention

### 4.2.c. Interventions

| Туре | Name | Description |
|---|---|---|
| Behavioral (e.g.,<br>Psychotherapy,<br>Lifestyle<br>Counseling) | Radicalizing Respect and Relationships (R3) | The theoretically grounded R3 Prevention Initiative (R3-PI) follows best practices for effective health behavior prevention programming, and is expected to include eight, 45-minute modules intended for delivery as an online synchronous program |

| 4.2.d. \$ | Study Phase | | Phase 1/2 | | |
|---|---|---|---|---|---|
| I | Is this an NIH-defined | Phase III Clinical Trial? | ○ Yes | <ul><li>No</li></ul> | |
| 4.2.e. l | Intervention Model | | Parallel | | |
| 4.2.f. N | Masking | | Yes | <ul><li>No</li></ul> | |
| | | □ Participant | ☐ Care Provider | ☐ Investigator | ☐ Outcomes Assessor |
| 4.2.g. / | Allocation | | Randomized | | |

#### 4.3. Outcome Measures

| Туре | Name | Time Frame | Brief Description |
|---|---|---|---|
| Primary | Alcohol Use | Past month at all time points | We will use the Timeline Followback to assess for alcohol use. |
| Primary | Dating Violence (Victimization and Perpetration) | Past 3 months (Baseline and 3-month follow-up); Past 1 month (immediate post-test) | We will use the Conflict in Adolescent Dating Relationships-Short Form and the Partner Cyber Abuse Questionnaire to assess for DV victimization and perpetration. |
| Secondary | Risky Sexual Behavior | Past 3 months (Baseline and 3-month follow-up); Past 1 month (immediate post-test) | We will use the Sexual Risk Survey to measure risky sexual behaviors. |

| Secondary | Depression | Past 3 months (Baseline and 3-month follow-up); Past 1 month (immediate post-test) | We will use the Kutcher Adolescent Depression Scale to measure depressive symptoms. |
|---|---|---|---|
| Secondary | Drug Use | Past 3 months (Baseline and 3-month follow-up); Past 1 month (immediate post-test) | We will us the Drug Use Disorders Identification Test to measure drug use. |
| Other | Identity Concealment (intermediary outcome) | N/A | We will use the Nebraska Outness Inventory to measure concealment of ones sexual identity. |
| Other | Internalized homonegativity (intermediary outcome) | N/A | We will use the Coming Out Self-efficacy Scale to measure internalized homonegativity |
| Other | Sense of LGBTQ+ Community (intermediary outcome) | N/A | We will use the Psychological Sense of LGBT Community Scale to measure sense of LGBTQ+ community. |
| Other | Healthy Coping (intermediary outcome) | N/A | We will use items adapted from Hamby et al.<br>Emotion Regulation Scale and the Drinking<br>Motives Questionnaire-Revised |
| Other | Conflict Resolution Skills (intermediary outcome) | N/A | We will use the Communication Skills & Response to Anger subscales to measure conflict resolution skills |
| Other | Refusal Skills (intermediary outcome) | N/A | We will use the Sexual Assertiveness Scale-W and the Drinking Refusal Self-Efficacy Questionnaire-Revised to measure refusal skills for sexual DV and alcohol, respectively. |
| Other | Bystander Behavior<br>(intermediary outcome) | N/A | We will use items adapted from Cook-Craig et al. (for DV) and items adapted from Oster-Aaland et al. and Krieger et al. (for AU) |
| Other | Social Norms (intermediary outcome) | N/A | We will use items adapted from the Readiness<br>to Help Scale- Denial Subscale (for DV) and<br>Drinking Norms Rating Form (for AU) |
| Other | Protective Behavioral<br>Strategies (intermediary<br>outcome) | N/A | We will use the Protective Behavioral Strategies Scale to measure protective behavioral strategies. |
| Secondary | Alcohol Consequences | Past month at all time points | We will use the Brief Young Adult Alcohol Consequences Questionnaire to assess for alcohol consequences. |

| 4.4. Statistical Design and Power | StatisticalDesignandPower_032020.pdf |
|-------------------------------------|--------------------------------------|
| 4.5. Subject Participation Duration | <1 year |

4.6.a. If yes, describe the availability of Investigational Product (IP) and Investigational New Drug (IND)/ Investigational Device Exemption (IDE) status

4.7. Dissemination Plan DisseminationPlan\_032020.pdf